CLINICAL TRIAL: NCT02949076
Title: Skeletal Muscle Atrophy and Dysfunction in Human Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: University of South Carolina (Other)
Responsible Party: Principal Investigator, Michael J. Toth, Ph.D., Associate Professor of Medicine, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16-506
Record Dates: First submitted 2016-10-25; First posted 2016-10-31 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise (Experimental): Lung cancer patients will undergo unilateral resistance exercise 3 times per week for 8 weeks during cancer treatment, while the other leg remains unexercised and will serve as a within-subject control.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Unilateral lower limb resistance exercise will be performed 3 times per week for 8 weeks in non-small cell lung cancer patients on only one leg, while the contralateral leg serves as a non-exercising control.

SUMMARY:
Cancer and its treatment can have profound effects on skeletal muscle, the most well-recognized being atrophy, weakness and diminished oxidative capacity. These adaptations negatively impact quality of life, treatment decisions and survival. Despite these consequences, the factors promoting these adaptations remain poorly defined and understudied in human patients. To address this gap in knowledge, our goal in this study is to examine the role of muscle disuse as a regulator of muscle size and function in human cancer patients

ELIGIBILITY:
Inclusion Criteria:

* 50-75 yrs of age
* histologically-documented, stage III or IV non-small cell lung carcinoma (NSCLC)
* estimated life expectancy >6 mos
* Karnofsky's performance score of ≥70

Exclusion Criteria:

* history, signs or symptoms of inflammatory or autoimmune disease
* uncontrolled hypertension
* heart or renal failure
* exercise limitations from peripheral vascular disease or stroke
* neuromuscular disease
* knee/hip replacement
* additional, actively-treated malignancy or history of malignancy, except non-melanoma skin cancer
* taking medication that can have anti-coagulant effects that cannot be stopped prior to the muscle biopsy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-07; Primary Completion 2023-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Cross-sectional area of skeletal muscle fibers | Difference between the change in the exercised and non-exercised leg from baseline to 8 weeks
  Cross-sectional area of skeletal muscle fibers will be evaluated using immunohistochemistry, with specification of all relevant muscle fiber types
Single muscle fiber contractile function | Difference between the change in the exercised and non-exercised leg from baseline to 8 weeks
  Segments of chemically-skinned single human muscle fibers will be assessed for cellular and molecular contractile parameters under maximal calcium-activated conditions, with muscle fiber type determined post-measurement by gel electrophoresis
Mitochondrial content | Difference between the change in the exercised and non-exercised leg from baseline to 8 weeks
  Mitochondrial content will be assessed by electron microscopy.
Mitochondrial function | Difference between the change in the exercised and non-exercised leg from baseline to 8 weeks
  Mitochondrial function will be assessed on isolated mitochondria

SECONDARY OUTCOMES:
Whole muscle size | Difference between the change in the exercised and non-exercised leg from baseline to 8 weeks
  Whole muscle size will be measured by computed tomography at the mid-thigh level.
Whole muscle isometric function | Difference between the change in the exercised and non-exercised leg from baseline to 8 weeks
  Whole muscle volitional contractile function will be measured by isometric Difference between the change in the exercised and non-exercised leg from baseline to 8 weeks by isometric dynamometry.
Whole muscle isokinetic function | Difference between the change in the exercised and non-exercised leg from baseline to 8 weeks
  Difference between the change in the exercised and non-exercised leg from baseline to 8 weeks by isokinetic dynamometry

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Toth, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- University of Vermont College of Medicine, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Yes
Research data (deidentified) which documents, supports and validates research findings will be stored on the University of Vermont College of Medicine computer system and will be made available upon final acceptance for publication of the major findings from the proposed studies. This includes raw data generated from all clinical and laboratory-based assessments under a data-sharing agreement.